CLINICAL TRIAL: NCT05396326
Title: Neoadjuvant Transcatheter Arterial Chemoinfusion and Embolism (TACiE) for Patients With Locally Advanced Adenocarcinoma of Stomach and Gastroesophageal Junction: a Pilot Study
Brief Title: A Pilot Study of Neoadjuvant TACiE in Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-TACiE01
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer
Keywords: neoadjuvant therapy; transcatheter arterial infusion; transcatheter arterial embolism; SOX
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; tegafur-gimeracil-oteracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX-TACiE (Experimental): Preoperative transcatheter arterial chemoinfusion and embolism (TACiE) alternated with systemic chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Teysuno; Procedure: Transarterial arterial chemoinfusion and embolism (TACiE)

INTERVENTIONS:
Drug: Oxaliplatin — The first and third cycles : transcatheter arterial infusion of oxaliplatin 85mg/m2, day 1.
  The second and fourth cycles: intra-venous oxaliplatin 135mg/m2, day 1.
Drug: Teysuno — Oral S-1, 40mg-60mg bid, day 1-14 for four 21-day cycles.
Procedure: Transarterial arterial chemoinfusion and embolism (TACiE) — In the first and third cycles : transcatheter arterial infusion of oxaliplatin 85mg/m2, day 1; transcatheter arterial embolism of tumor feeding arteries, day 1, if applicable.

SUMMARY:
This is a prospective pilot study to evaluate the safety and feasibility of neoadjuvant transcatheter infusion and embolism (TACiE) in patients with locally advanced adenocarcinoma of stomach and gastroesophageal junction.

The TACiE protocol includes four cycles. Transcatheter oxaliplatin and concurrent embolism on day 1 and oral S-1 on day 1-14 will be administrated in the first and third cycles. Intra-venous oxaliplatin on day 1 and oral S-1 on day 1-14 (SOX) will be administrated in the second and fourth cycles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years old;
* The Karnofsky Performance Scale (KPS) score >=80;
* Adenocarcinoma of stomach and gastroesophageal junction (Siewert II/III) diagnosed pathologically;
* clinical T3-4a/N+/M0 (The 8th edition of the American Joint Committee on Cancer (AJCC) staging system);
* According to the Response Evaluation Criteria In Solid Tumours (RECIST) 1.1 standard, there is at least one evaluable lesion in the abdominal CT/MRI;
* The surgeons participating in this study judged the lesion to be resectable;
* Physical condition allows the surgery;

Exclusion Criteria:

* Distant metastasis or local unresectable factors;
* Cytotoxic chemotherapy, radiotherapy, immunotherapy or radical surgery for the treatment of this gastric cancer, except for corticosteroids;
* Active autoimmune diseases or a history of autoimmune diseases;
* History of malignant tumors within 2 years;
* Gastrointestinal bleeding within two weeks prior to enrollment, or those with high bleeding risk;
* Gastrointestinal perforation and/or fistula occurred within 6 months before enrollment;
* Upper gastrointestinal obstruction or abnormal physiological function or suffering from malabsorption syndrome, which may affect the absorption of drugs;
* Weight loss >=20% within 2 months before enrollment;
* A history of the following lung diseases: interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, etc.;
* Uncontrollable systemic diseases including diabetes, hypertension, etc.; Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis, HIV infection, etc.;
* Untreated patients with chronic hepatitis B or chronic HBV carriers with hepatitis B virus (HBV) DNA exceeding 500 IU/mL, or hepatitis C virus (HCV) RNA positive patients should be excluded;
* Any of the following cardiovascular risk factors (refer to Research Guide);
* Known peripheral nerve disease >=NCI CTCAE Grade 1. However, patients with only the disappearance of the deep tendon reflex (DTR) need not be excluded;
* Moderate or severe renal damage [creatinine clearance equal to or lower than 50 ml/min (calculated according to the Cockcroft and Gault equation)], or serum creatinine> upper limit of normal (ULN); People with known dihydropyrimidine dehydrogenase (DPD) deficiency;
* Those who are allergic to any research drug ingredients;
* Underwent major surgery within 28 days prior to enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment related adverse events (TRAE). | up to 28 days after last dose of preoperative therapy
  The percentage of patients who developed TRAE

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | two weeks after surgery
  The percentage of patients found no tumor residual in primary tumor and resected lymph nodes.
Objective response rate (ORR) | up to 3 months
  The percentage of patients found complete response or partial response to preoperative therapy according to RECIST v1.1.
Overall survival (OS) | From date of enrollment until the date of death from any cause, assessed up to 36 months
  The time from enrollment to death caused by any causes or censor.
Progressive free survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The time from enrollment to tumor progression, death or censor.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- [Background] Sasako M, Sano T, Yamamoto S, Sairenji M, Arai K, Kinoshita T, Nashimoto A, Hiratsuka M; Japan Clinical Oncology Group (JCOG9502). Left thoracoabdominal approach versus abdominal-transhiatal approach for gastric cancer of the cardia or subcardia: a randomised controlled trial. Lancet Oncol. 2006 Aug;7(8):644-51. doi: 10.1016/S1470-2045(06)70766-5. PMID 16887481
- [Background] Sano T, Sasako M, Mizusawa J, Yamamoto S, Katai H, Yoshikawa T, Nashimoto A, Ito S, Kaji M, Imamura H, Fukushima N, Fujitani K; Stomach Cancer Study Group of the Japan Clinical Oncology Group. Randomized Controlled Trial to Evaluate Splenectomy in Total Gastrectomy for Proximal Gastric Carcinoma. Ann Surg. 2017 Feb;265(2):277-283. doi: 10.1097/SLA.0000000000001814. PMID 27280511
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Schuhmacher C, Gretschel S, Lordick F, Reichardt P, Hohenberger W, Eisenberger CF, Haag C, Mauer ME, Hasan B, Welch J, Ott K, Hoelscher A, Schneider PM, Bechstein W, Wilke H, Lutz MP, Nordlinger B, Van Cutsem E, Siewert JR, Schlag PM. Neoadjuvant chemotherapy compared with surgery alone for locally advanced cancer of the stomach and cardia: European Organisation for Research and Treatment of Cancer randomized trial 40954. J Clin Oncol. 2010 Dec 10;28(35):5210-8. doi: 10.1200/JCO.2009.26.6114. Epub 2010 Nov 8. PMID 21060024
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Al-Batran SE, Homann N, Pauligk C, Goetze TO, Meiler J, Kasper S, Kopp HG, Mayer F, Haag GM, Luley K, Lindig U, Schmiegel W, Pohl M, Stoehlmacher J, Folprecht G, Probst S, Prasnikar N, Fischbach W, Mahlberg R, Trojan J, Koenigsmann M, Martens UM, Thuss-Patience P, Egger M, Block A, Heinemann V, Illerhaus G, Moehler M, Schenk M, Kullmann F, Behringer DM, Heike M, Pink D, Teschendorf C, Lohr C, Bernhard H, Schuch G, Rethwisch V, von Weikersthal LF, Hartmann JT, Kneba M, Daum S, Schulmann K, Weniger J, Belle S, Gaiser T, Oduncu FS, Guntner M, Hozaeel W, Reichart A, Jager E, Kraus T, Monig S, Bechstein WO, Schuler M, Schmalenberg H, Hofheinz RD; FLOT4-AIO Investigators. Perioperative chemotherapy with fluorouracil plus leucovorin, oxaliplatin, and docetaxel versus fluorouracil or capecitabine plus cisplatin and epirubicin for locally advanced, resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4): a randomised, phase 2/3 trial. Lancet. 2019 May 11;393(10184):1948-1957. doi: 10.1016/S0140-6736(18)32557-1. Epub 2019 Apr 11. PMID 30982686
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Smalley SR, Benedetti JK, Haller DG, Hundahl SA, Estes NC, Ajani JA, Gunderson LL, Goldman B, Martenson JA, Jessup JM, Stemmermann GN, Blanke CD, Macdonald JS. Updated analysis of SWOG-directed intergroup study 0116: a phase III trial of adjuvant radiochemotherapy versus observation after curative gastric cancer resection. J Clin Oncol. 2012 Jul 1;30(19):2327-33. doi: 10.1200/JCO.2011.36.7136. Epub 2012 May 14. PMID 22585691
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- [Background] Su Z, Shu K, Kang M, Wang G. Pathological complete response from oral chemotherapy combined with trans-arterial chemotherapy and embolization in an unresectable gastric cancer patient: A case report. Medicine (Baltimore). 2019 Jun;98(25):e16075. doi: 10.1097/MD.0000000000016075. PMID 31232946